CLINICAL TRIAL: NCT03370094
Title: Prehospital Identification of Patients With Suspected Stroke Using Onsite Mobile Telemedicine
Brief Title: Tele-Stroke: Prehospital Identification of Patients With Suspected Stroke Using Onsite Mobile Telemedicine - Feasibility
Acronym: Tele-Stroke
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: propatient Basel (Unknown)
Responsible Party: Sponsor
Other Study IDs: PP-16-23
Record Dates: First submitted 2017-11-28; First posted 2017-12-12 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with suspected stroke: patients with suspected stroke due to paramedic's initial evaluation of face, arm, and speech function will be diagnosed with audio-video-streaming of suspected stroke symptoms and signs
  Interventions: Diagnostic Test: Audio-video-streaming of suspected stroke symptoms and signs

INTERVENTIONS:
Diagnostic Test: Audio-video-streaming of suspected stroke symptoms and signs — The diagnosis based on the patient evaluation by end-to-end encrypted real-time video will be compared to the gold standard, consisting of an in-person neurological examination by a stroke specialist in patients with suspected acute stroke.

SUMMARY:
Observational Study to investigate the technical feasibility, implementation into current diagnostic and treatment pathways and the diagnostic accuracy of the remote patient assessment by using mobile telecommunication ahead of hospitalization.

DETAILED DESCRIPTION:
On-site, pre-hospital clinical assessment of patients with suspected acute stroke can accelerate further diagnostic and treatment pathways after patient arrival at the emergency room or the dedicated stroke center. Interactive video and audio streaming connecting on-site paramedics to a stroke center based stroke physicians can help to overcome these hurdles. Patient evaluation by simple, pre-defined assessment measures and a standardized questionnaire may enable a pre-hospital decision on the need of expedited diagnostic and treatment procedures after arrival at the dedicated stroke center.

ELIGIBILITY:
Inclusion Criteria:

* Any patient older or equal than 18 years with suspected acute stroke as per the first judgement of the paramedics on-site.
* written informed consent by the patient, or legal representative (next-of kin) or informed consent by an independent physician not involved in the study

Exclusion Criteria:

-patients with symptoms not attributable to stroke in the emergency onsite ( observation of epileptic seizure, recent cerebral trauma, prior syncope or comatose state)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The current phase of the project ("Feasibility") will include patients with suspected acute stroke already admitted to the ER of the University Hospital Basel, and patients with suspected acute stroke and who are referred to the Stroke Center of USB by the paramedics.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the patient evaluation by remote Audio/video session | 1 hour
  The proportion of successfully realized 'telestroke' interviews (=patient has a stroke yes/no) in comparison to final diagnosis by the caring stroke team.

SECONDARY OUTCOMES:
Diagnostic accuracy of an automated biometric software | 12 months
  The proportion of correct stroke diagnosis by the automatic biometric assessment compared to the final diagnosis of the caring stroke team.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lyrer, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No